CLINICAL TRIAL: NCT04441996
Title: Therapeutic Plasma Exchange for COVID-19-associated Hyperviscosity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Cheryl Maier, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000949
Record Dates: First submitted 2020-06-19; First posted 2020-06-22 (Actual); Results first posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-11

CONDITIONS: COVID-19
Keywords: Hyperviscosity
MeSH Terms: conditions — COVID-19; Thrombophilia | interventions — Plasma Exchange; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Therapeutic plasma exchange (TPE) (Experimental): Participants with COVID-19-associated hyperviscosity randomized to receive therapeutic plasma exchange (TPE).
  Interventions: Biological: Therapeutic plasma exchange (TPE)
- Standard of care (Active Comparator): Participants with COVID-19-associated hyperviscosity randomized to receive standard of care treatment.
  Interventions: Other: Standard of care

INTERVENTIONS:
Biological: Therapeutic plasma exchange (TPE) — Participants will receive two treatments of TPE with frozen plasma (FP) replacement on two sequential days (Day 2 and Day 3). All procedures will be performed by the apheresis staff at the hospital sites, following institutional standard operating procedures. FP will be obtained from American Red Cross or LifeSouth Community Blood centers.
  Arms: Therapeutic plasma exchange (TPE)
Other: Standard of care — Participants will continue to receive standard of care and be closely monitored by ICU team for any change in clinical status, and any adverse events directly related to study intervention will be reported to the study investigator.
  Arms: Standard of care

SUMMARY:
Many patients with Coronavirus Disease 2019 (COVID-19) have atypical blood clots. These blood clots can occur in either veins or arteries and be large, like in stroke or heart attack, or very tiny, called microthrombi. Some patients with COVID-19 even have blood clots despite being on anti-clotting medications. Blood with increased viscosity does not flow through the body normally, in the same way that syrup, a highly viscous liquid, and water, a minimally viscous liquid, flow differently. The researchers believe that hyperviscosity may contribute to blood clots and organ damage seen in patients with severe COVID-19. Plasma exchange removes a patient's plasma, which contains the large sticky factors that the researchers believe are increasing viscosity, and replaces it with plasma from healthy donors. In addition to providing important information about plasma exchange as a treatment in COVID-19 for patients, this study will provide data to justify resource and staffing decisions.

This study will enroll 20 participants who are critically ill from COVID-19. Participants will be randomized to receive therapeutic plasma exchange (TPE) or standard of care (SOC).

DETAILED DESCRIPTION:
Critically ill COVID-19 patients have high rates of complications, including respiratory failure, renal impairment, and a coagulopathic state that may exacerbate these conditions and contribute to additional end organ injury. Consistent with a fundamentally distinct nature of COVID-19-associated disease, our preliminary studies demonstrate that patients with COVID-19 exhibit an increase in plasma viscosity. Furthermore, the researchers have found that plasma viscosity strongly correlates with sequential organ failure assessment (SOFA) scores, a mortality prediction score used in the intensive care unit (ICU), in COVID-19 infected patients. These results strongly suggest that altered blood flow secondary to hyperviscosity may contribute to end organ injury and therefore morbidity and mortality in the most critically ill COVID-19 patients. More detailed analysis of the potential etiology of COVID-19-associated plasma hyperviscosity has demonstrated that these patients also have significantly elevated levels of the plasma protein fibrinogen. Increased fibrinogen levels, which may be either entirely responsible for or at least contribute to hyperviscosity in these patients, may be the primary mediator of refractory hypercoagulability in this patient population. Thus, hyperviscosity induced by hyperfibrinogenemia may be a critical driver of morbidity and mortality in patients with COVID-19.

Therapeutic plasma exchange (TPE) is the only procedure known to directly and rapidly decrease plasma viscosity, suggesting that TPE may improve patient outcomes in critically ill patients with COVID-19 by decreasing plasma viscosity and thereby enhancing blood flow. However, as a procedure, extensive implementation of TPE would require significant devotion of hospital resources, including apheresis machines and the staff needed to successfully conduct these procedures. The procedures alone require staff to have prolonged interactions with critically ill COVID-19 patients, placing them at a potentially increased risk for contracting COVID-19. It is therefore essential that clear and unequivocal data be generated in order to accurately assess the risk and benefits of this procedure for both patients and staff. Such data will also aid in determining the necessary resources that may be needed to successfully conduct TPE for this patient population.

Participants will be randomized in a 1:1 ratio to receive TPE or SOC. Participants in the TPE study arm will receive two treatments of TPE with frozen plasma on sequential days. Plasma viscosity will be measured before TPE (Day 1) and following the second TPE treatment (Day 3 or 4). Participants in the SOC study arm will also have their plasma viscosity assessed on Days 1 and 3. Participants will be followed for the duration of their hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients admitted to the ICU at Emory University Hospital, Emory University Hospital Midtown, or Emory Saint Joseph's Hospital
* Evidence of COVID-19 infection documented by a laboratory test either by one of the following:

  * A diagnostic test (e.g., nasopharyngeal swab, tracheal aspirate, other)
  * Positive serological test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) antibodies
  * Medical records from outside institution
* Plasma viscosity >2.3 and <3.5 centipoise (cp) or Fibrinogen >800 mg/dL

Exclusion Criteria:

* Patients with plasma viscosity > 3.5 cp
* Moribund patients that the ICU clinical team expects to die within 24 hours
* Patients with any condition that, in the opinion of the clinical team or investigator, could increase the subject's risk by participating in the study or confound the outcome of the study
* Patients participating in another clinical trial that prohibits the use of TPE
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Maier, MD, PhD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Emory University Hospital, Emory University Hospital Midtown, and Emory Saint Joseph's Hospital in Atlanta, Georgia, USA. Participant enrollment began July 17, 2020 and all follow-up assessments were completed by March 18, 2021.
Groups:
- Therapeutic Plasma Exchange (TPE): Participants with Coronavirus Disease 2019 (COVID-19) associated elevated plasma viscosity randomized to receive therapeutic plasma exchange (TPE) with frozen plasma. Participants were randomized on Day 1 and received two treatments of TPE on sequential days (Day 2 and Day 3).
- Standard of Care: Participants with COVID-19-associated elevated plasma viscosity randomized to receive standard of care treatment.
Period: Overall Study
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Therapeutic Plasma Exchange (TPE): Participants with COVID-19-associated elevated plasma viscosity randomized to receive therapeutic plasma exchange (TPE) with frozen plasma. Participants were randomized on Day 1 and received two treatments of TPE on sequential days (Day 2 and Day 3).
- Total: Total of all reporting groups
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (14.4) | 58.8 (9.04) | 58.9 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 9 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 7 | 12
  Unknown or Not Reported | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 5 | 12
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Plasma Viscosity
Description: Plasma viscosity is measured in centipoise (cP). The normal range is 1.4 - 1.8 cP and measurements above this range indicate increased viscosity.
Time Frame: Day 1 (within 24 hours prior to TPE), Day 4 (within 24 hours of last TPE)
Measure: Mean (Standard Deviation); unit: cP
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 10 | 10
cP
  Baseline | 2.35 (0.37) | 2.47 (0.34)
  Post-treatment | 1.61 (0.09) | 2.47 (0.48)

2. Primary Outcome: Cumulative Incidence of Adverse Events
Description: The primary safety endpoint is assessed as the cumulative incidence of adverse events directly associated with TPE during the study period as determined by clinical judgment of ICU team providing direct patient care and the study PI.
Time Frame: Up to Day 28
Population: This analysis includes participants in the TPE study arm.
Measure: Number; unit: adverse events
Arm/Group | Therapeutic Plasma Exchange (TPE)
Number analyzed (Participants) | 10
adverse events | 1

3. Secondary Outcome: Cumulative All Cause Mortality
Description: The number of participants dying from any cause is reported as a cumulative measures of mortality.
Time Frame: Up to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 10 | 10
Participants
  Day 1 to Day 3 | 0 | 0
  Day 1 to Day 7 | 0 | 0
  Day 1 to Day 14 | 0 | 2
  Day 1 to Day 21 | 1 | 4
  Day 1 to Day 28 | 2 | 5

4. Secondary Outcome: Cumulative Count of Bleeding and Thromboembolic Complications
Description: The number of bleeding and thromboembolic complications will be compared between study arms. This endpoint is a composite outcome including any acute bleeding requiring transfusion support, venous thrombosis (deep vein thrombosis or pulmonary embolism), arterial clots (myocardial infarction, stroke, limb ischemia), renal replacement therapy or catheter line related clots. The values reported are cumulative.
Time Frame: Up to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 10 | 10
Participants
  Day 1 to Day 3 | 0 | 0
  Day 1 to Day 7 | 1 | 0
  Day 1 to Day 14 | 1 | 0
  Day 1 to Day 21 | 2 | 2
  Day 1 to Day 28 | 2 | 2

5. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure will be assessed in days and is defined as plasma viscosity > 3.5 cP and/or the participant is offered TPE outside of trial by primary clinical team.
Time Frame: Up to Day 28
Population: This analysis includes participants experiencing treatment failure.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 2 | 2
days | 5.5 (2.12) | 2.5 (3.54)

6. Secondary Outcome: Duration of ICU Stay
Description: The number of days spent in the ICU after study enrollment is presented here. All patients are included in calculating the reported mean, including those whose ICU stay ended due to death.
Time Frame: Up to Day 48
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 10 | 10
days | 23.1 (15.7) | 16.0 (11.4)

7. Secondary Outcome: Duration of Hospital Stay
Description: The number of days spent hospitalized after study enrollment is presented here. All patients are included in calculating the reported mean, including those whose hospitalization ended due to death.
Time Frame: Up to Day 48
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 10 | 10
days | 27.2 (12.4) | 21.7 (12.0)

8. Secondary Outcome: Discharge Disposition
Description: The number of participants in each study arm discharged to home or to a long-term acute care (LTAC) hospital, versus palliative care or death.
Time Frame: Up to Day 48
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 10 | 10
Participants
  Home or LTAC | 7 | 5
  Palliative care or death | 3 | 5

9. Secondary Outcome: Clinical Status Score
Description: The clinical status of participants was assessed using a single item modified from the World Health Organization (WHO) ordinal clinical severity scale for COVID. The instrument was customized for this study to evaluate thrombotic/bleeding events. In this 12-point ordinal scale, a score of 1 indicates no evidence of infection and the severity of the clinical status increases as the number of necessary interventions increases to the final score of 12, which is death. All patients were included at every timepoint recorded, with "terminal" scores carried over from the measure before for those that expired or fully recovered.
Time Frame: Day 1 (day of study enrollment), Day 4 (one day after second TPE treatment), Days 7, 14, 21, and 28
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 10 | 10
score on a scale
  Day 1 (day of study enrollment) | 7.0 [6.0 to 7.75] | 8.0 [7.25 to 8.0]
  Day 4 (1 day after second TPE treatment) | 7.0 [6.0 to 7.0] | 8.0 [7.25 to 8.0]
  Day 7 | 7.0 [6.0 to 8.0] | 8.0 [7.0 to 8.0]
  Day 14 | 8.0 [6.0 to 8.0] | 7.5 [7.0 to 9.75]
  Day 21 | 7.5 [5.5 to 8.0] | 8.0 [7.0 to 12.0]
  Day 28 | 7.0 [5.5 to 8.75] | 10.0 [7.0 to 12.0]

10. Secondary Outcome: Body Temperature
Description: Body temperature will be assessed in degrees Celsius.
Time Frame: Days 7, 14, 21, and 28
Population: Body temperature was not collected in an effort to reduce redundancy and workload for clinicians as more relevant/direct measures were already being collected.
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure will be assessed in millimeters of mercury (mm Hg).
Time Frame: Days 7, 14, 21, and 28
Population: Blood pressure was not collected in an effort to reduce redundancy and workload for clinicians as more relevant/direct measures were already being collected.
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Diastolic Blood Pressure
Description: Diastolic blood pressure will be assessed in millimeters of mercury (mm Hg).
Time Frame: Days 7, 14, 21, and 28
Population: as for outcome 11
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Heart Rate
Description: Heart rate will be assessed as beats per minute.
Time Frame: Days 7, 14, 21, and 28
Population: Heart rate was not collected in an effort to reduce redundancy and workload for clinicians as more relevant/direct measures were already being collected.
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Respiratory Rate
Description: Respiratory rate will be assessed as breaths per minute.
Time Frame: Days 7, 14, 21, and 28
Population: Respiratory rate was not collected in an effort to reduce redundancy and workload for clinicians as more relevant/direct measures were already being collected.
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Ventilator Days
Description: The number of days participants are on a ventilator, among participants who were ever on a ventilator after study enrollment.
Time Frame: Up to Day 28
Population: This analysis includes participants who were on a ventilator; two participants in the TPE arm were never on a ventilator.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 8 | 10
days | 22.6 (11.6) | 19.2 (11.2)

16. Secondary Outcome: Ventilator Oxygen Percent (FiO2)
Description: The oxygen percent delivered with a ventilator that is needed to maintain blood oxygen levels will be compared between study arms.
Time Frame: Days 7, 14, 21, and 28
Population: FiO2 was not collected in an effort to reduce redundancy and workload for clinicians as more relevant/direct measures were already being collected.
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Positive End-Expiratory Pressure (PEEP)
Description: PEEP during ventilator use is measured in centimeters of water (cmH2O) and is the pressure in the lungs above atmospheric pressure, at the end of an exhalation. Higher PEEP (10 cmH2O or greater) may be associated with improved mortality, compared with PEEP below 10 cmH2O.
Time Frame: Day 1 (day of study enrollment), Day 4 (one day after second TPE treatment), Days 7, 14, 21, and 28
Population: This analysis includes participants who were assessed for PEEP at the indicated time point.
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 5 | 7
cmH2O
  Day 1 (day of study enrollment): number analyzed (Participants) | 3 | 7
  Day 1 (day of study enrollment) | 12.7 (5.0) | 15.9 (5.9)
  Day 4 (one day after second TPE treatment): number analyzed (Participants) | 5 | 6
  Day 4 (one day after second TPE treatment) | 11.6 (4.3) | 13.0 (3.7)
  Day 7: number analyzed (Participants) | 4 | 6
  Day 7 | 13.0 (6.2) | 11.3 (3.9)
  Day 14: number analyzed (Participants) | 4 | 6
  Day 14 | 13.0 (2.0) | 13.3 (2.7)
  Day 21: number analyzed (Participants) | 4 | 4
  Day 21 | 11.0 (1.2) | 11.0 (2.0)
  Day 28: number analyzed (Participants) | 4 | 3
  Day 28 | 11.0 (2.6) | 12.7 (7.0)

18. Secondary Outcome: Vasopressor Requirements
Description: Whether or not breathing assistance from vasopressors is needed will be compared between study arms.
Time Frame: Days 7, 14, 21, and 28
Population: Vasopressor requirements were not collected in an effort to reduce redundancy and workload for clinicians as more relevant/direct measures were already being collected.
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Need for Treatment From a Registered Respiratory Therapist (RRT)
Description: Whether or not breathing assistance from an RRT is needed will be compared between study arms.
Time Frame: Days 7, 14, 21, and 28
Population: Need for treatment from an RRT was not collected in an effort to reduce redundancy and workload for clinicians as more relevant/direct measures were already being collected.
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Sequential Organ Failure Assessment (SOFA) Score
Description: The Sequential Organ Failure Assessment (SOFA) score is a method of predicting mortality that is based on the degree of dysfunction of six organ systems (respiratory, nervous, cardiovascular, liver, coagulation, and kidneys). Each organ system is scored between 0 and 4, where 0 indicates normal function and 4 indicates a high degree of dysfunction. Total scores range from 0 to 24. A score of 0-6 is associated with a mortality rate of less than 10% while a score between 16 and 24 is associated with a greater than 90% mortality rate.
Time Frame: Day 1 (day of study enrollment), Day 4 (one day after second TPE treatment), Days 7, 14, 21, and 28
Population: This analysis includes participants who had a SOFA score assessment at the indicated time point.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 10 | 10
score on a scale
  Day 1 (day of study enrollment) | 10.5 [8.5 to 12.75] | 13.0 [11.25 to 14.0]
  Day 4 (one day after second TPE treatment) | 11.0 [7.75 to 12.5] | 11.5 [11.0 to 12.75]
  Day 7 | 11.0 [10.0 to 12.0] | 12.0 [11.25 to 13.75]
  Day 14 | 12.5 [8.75 to 13.75] | 12.5 [11.0 to 15.0]
  Day 21: number analyzed (Participants) | 9 | 8
  Day 21 | 11.5 [8.75 to 12.0] | 13.0 [10.75 to 15.75]
  Day 28: number analyzed (Participants) | 7 | 4
  Day 28 | 11.5 [8.25 to 12.75] | 12.0 [9.0 to 15.75]

21. Secondary Outcome: Partial Pressure of Arterial Oxygen (PaO2)/Percentage of Inspired Oxygen (FiO2) Ratio
Description: The PaO2/FiO2 ratio is decreased with hypoxia. A value of less than 200 indicates acute respiratory distress syndrome (ARDS).
Time Frame: Day 1 (day of study enrollment), Day 4 (one day after second TPE treatment), Days 7, 14, 21, and 28
Population: This analysis includes participants with available arterial blood gas (ABG) values.
Measure: Mean (Standard Deviation); unit: PaO2/FiO2 ratio
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 5 | 9
PaO2/FiO2 ratio
  Day 1 (day of study enrollment): number analyzed (Participants) | 5 | 8
  Day 1 (day of study enrollment) | 219 (102) | 166 (79)
  Day 4 (one day after second TPE treatment) | 132 (80) | 157 (44)
  Day 7: number analyzed (Participants) | 5 | 6
  Day 7 | 151 (131) | 141 (54)
  Day 14: number analyzed (Participants) | 5 | 5
  Day 14 | 109 (21) | 101 (43)
  Day 21: number analyzed (Participants) | 5 | 2
  Day 21 | 104 (32) | 145 (2)
  Day 28: number analyzed (Participants) | 3 | 2
  Day 28 | 108 (54) | 146 (127)

22. Secondary Outcome: Ventilatory Ratio
Description: Ventilatory ratio will be documented. The formula for the ventilatory is [minute ventilation (ml/min) × PaCO2 (mm Hg)]/(predicted body weight × 100 × 37.5).
Time Frame: Days 7, 14, 21, and 28
Population: Information for calculating the ventilatory ratio was not collected in an effort to reduce redundancy and workload for clinicians as more relevant/direct measures were already being collected.
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: White Blood Count (WBC)
Description: The normal range for WBC is 3,400 to 6,600 cells per microliter (cells/mL) of blood. A high WBC occurs when inflammation or infection is present.
Time Frame: Days 7, 14, 21, and 28
Population: Information for this outcome was not collected for any participants. Limited laboratory data was available for clinical parameters ordered by the patients' healthcare providers as part of routine clinical care and later abstracted by study team members by chart review. This analyte was not abstracted by the study team for any patient given realization that too few points were available for analysis to generate meaningful data for interpretation.
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Hemoglobin (Hb)
Description: Hemoglobin is measured in grams per deciliter (grams/dL). A normal Hb count for males is 13.2 to 16.6 grams/dL and a normal count for females is 11.6 to 15 grams/dL. A patient has anemia when their hemoglobin is low.
Time Frame: Days 7, 14, 21, and 28
Population: as for outcome 23
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Hematocrit (Hct)
Description: A measure of hematocrit is the volume of red blood cells in the total blood volume. Normal hematocrit for males is 40 to 54% and a normal measurement for females is 36 to 48%
Time Frame: Days 7, 14, 21, and 28
Population: as for outcome 23
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Platelet Count
Description: A normal platelet is 150,000 to 450,000 platelets per microliter of blood. An excess of platelets in the blood can be caused by inflammation or infection.
Time Frame: Days 7, 14, 21, and 28
Population: as for outcome 23
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Mean Platelet Volume (MVP)
Description: MVP is a measurement of platelet size. Platelet size tends to be increased when platelet count is high. Typical platelet volume is 9.4 to 12.3 femtoliters (fL).
Time Frame: Days 7, 14, 21, and 28
Population: as for outcome 23
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Blood Urea Nitrogen (BUN)
Description: The normal range for BUN is 7 to 20 milligrams per deciliter (mg/dL) of blood. A high BUN value indicates that kidneys are not functioning well.
Time Frame: Days 7, 14, 21, and 28
Population: as for outcome 23
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Creatinine
Description: The normal range for creatinine is 0.84 to 1.21 mg/dL of blood. High serum creatinine indicates that kidneys are not functioning well.
Time Frame: Day 1 (day of study enrollment), Day 4 (one day after second TPE treatment), Days 7, 14, 21, and 28
Population: This analysis includes participants who had creatinine assessed at the indicated time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 10 | 10
mg/dL
  Day 1 (day of study enrollment) | 2.5 (2.1) | 2.9 (1.8)
  Day 4 (one day after second TPE treatment) | 2.0 (1.3) | 2.6 (1.7)
  Day 1: number analyzed (Participants) | 9 | 8
  Day 1 | 2.3 (1.4) | 2.6 (1.7)
  Day 14: number analyzed (Participants) | 9 | 8
  Day 14 | 2.6 (2.3) | 2.7 (1.8)
  Day 21: number analyzed (Participants) | 8 | 7
  Day 21 | 2.3 (3.3) | 2.8 (1.7)
  Day 28: number analyzed (Participants) | 6 | 4
  Day 28 | 1.3 (1.6) | 2.0 (1.6)

30. Secondary Outcome: Bilirubin
Description: For adults, normal values for total bilirubin are around 1.2 mg/dL of blood. High bilirubin indicates that the liver is not functioning well.
Time Frame: Days 7, 14, 21, and 28
Population: as for outcome 23
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 0 | 0

31. Secondary Outcome: Total Protein
Description: The normal range for total protein is 6.0 to 8.3 g/dL of blood. High levels of total protein can occur with inflammation or infection while low levels may indicate kidney or liver problems, or malnutrition.
Time Frame: Days 7, 14, 21, and 28
Population: as for outcome 23
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 0 | 0

32. Secondary Outcome: Albumin
Description: The normal range for albumin is 3.4 to 5.4 g/dL of blood. High albumin may indicate acute infection while low albumin can indicate malnutrition or liver disease.
Time Frame: Days 7, 14, 21, and 28
Population: as for outcome 23
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 0 | 0

33. Secondary Outcome: C-reactive Protein (CRP)
Description: A normal value for CRP (with a standard test) is less than 10 milligrams per liter (mg/L) of blood. CRP increases with inflammation, which could be attributed to an infection, chronic inflammatory disease or heart disease.
Time Frame: Day 1 (day of study enrollment), Day 4 (one day after second TPE treatment), Days 7, 14, 21, and 28
Population: This analysis includes participants who had CRP assessed at the indicated time point.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 10 | 10
mg/L
  Day 1 (day of study enrollment) | 226 (74) | 234 (115)
  Day 4 (one day after second TPE treatment) | 83 (37) | 179 (115)
  Day 7: number analyzed (Participants) | 9 | 6
  Day 7 | 153 (153) | 210 (91)
  Day 14: number analyzed (Participants) | 7 | 5
  Day 14 | 119 (94) | 195 (81)
  Day 21: number analyzed (Participants) | 7 | 2
  Day 21 | 149 (134) | 71 (27)
  Day 28: number analyzed (Participants) | 3 | 1
  Day 28 | 215 (213) | 141 (0)

34. Secondary Outcome: Interleukin 6 (IL-6)
Description: A normal value for IL-6 is 1.8 picograms per milliliter (pg/mL) or less. IL-6 is increased in patients with infections or chronic inflammation.
Time Frame: Days 7, 14, 21, and 28
Population: as for outcome 23
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 0 | 0

35. Secondary Outcome: Prothrombin Time (PT)
Description: Prothrombin time is a measurement of the time it takes (in seconds) for blood to clot. A normal value is 10 to 14 seconds.
Time Frame: Days 7, 14, 21, and 28
Population: as for outcome 23
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 0 | 0

36. Secondary Outcome: International Normalized Ratio (INR)
Description: An INR of around 1.1 is considered normal. Lower INR can means that blood is clotting faster than desired while higher INR indicates that blood is clotting slower than normal.
Time Frame: Days 7, 14, 21, and 28
Population: as for outcome 23
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 0 | 0

37. Secondary Outcome: Activated Partial Thromboplastin Time (aPTT)
Description: The aPTT test is a measurement of blood clotting time. Normal values for aPTT are around 30 to 40 seconds. Higher aPTT values can indicate a bleeding risk.
Time Frame: Days 7, 14, 21, and 28
Population: as for outcome 23
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 0 | 0

38. Secondary Outcome: Anti-factor Xa (Anti-Xa)
Description: The anti-factor Xa assay measures plasma heparin and is useful with monitoring anticoagulation therapy. Interpretation of the resulting values depends on the anticoagulation medication used as well as the dosing schedule and indication. Patients not taking heparin should have an anti-Xa value of 0 units per milliliter (U/mL).
Time Frame: Days 7, 14, 21, and 28
Population: as for outcome 23
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 0 | 0

39. Secondary Outcome: Fibrinogen
Description: Fibrinogen is a protein that helps with the formation of blood clots. For adults, the normal range of fibrinogen is 200 to 400 mg/dL. Fibrinogen can be increased in patients with liver, kidney, or inflammatory diseases. The risk of developing a thromboembolism is increased with chronically high levels of fibrinogen.
Time Frame: Day 1 (day of study enrollment), Day 4 (one day after second TPE treatment), Days 7, 14, 21, and 28
Population: This analysis includes participants who had fibrinogen assessed at the indicated time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 10 | 10
mg/dL
  Day 1 (day of study enrollment) | 934 (79) | 860 (182)
  Day 4 (one day after second TPE treatment) | 359 (71) | 807 (199)
  Day 7: number analyzed (Participants) | 7 | 5
  Day 7 | 663 (166) | 806 (189)
  Day 14: number analyzed (Participants) | 6 | 4
  Day 14 | 593 (143) | 762 (145)
  Day 21: number analyzed (Participants) | 7 | 3
  Day 21 | 687 (125) | 598 (89)
  Day 28: number analyzed (Participants) | 3 | 1
  Day 28 | 693 (33) | 116 (0)

40. Secondary Outcome: D-dimer
Description: The D-dimer blood test is a method of screening for deep vein thrombosis or pulmonary embolism. A normal D-dimer value is less than 0.50 micrograms per milliliter (mcg/mL) of blood. High levels of D-dimer can occur when a patient has a major blood clot, infection, or liver disease.
Time Frame: Day 1 (day of study enrollment), Day 4 (one day after second TPE treatment), Days 7, 14, 21, and 28
Population: This analysis includes participants who had D-dimer at the indicated time point.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
Number analyzed (Participants) | 10 | 10
mcg/mL
  Day 1 (day of study enrollment) | 5187 (8973) | 1632 (1163)
  Day 4 (one day after second TPE treatment) | 3519 (5575) | 6253 (9325)
  Day 7: number analyzed (Participants) | 9 | 7
  Day 7 | 4041 (6408) | 1749 (1126)
  Day 14: number analyzed (Participants) | 7 | 5
  Day 14 | 1819 (650) | 6767 (8304)
  Day 21: number analyzed (Participants) | 8 | 3
  Day 21 | 6765 (13044) | 3136 (1911)
  Day 28: number analyzed (Participants) | 4 | 1
  Day 28 | 16648 (28942) | 6567 (0)

ADVERSE EVENTS:
Time Frame: Information on TPE-associated adverse events was collected in patients receiving the study intervention (TPE) beginning with the initiation of the first TPE and continued up to 28 days after study enrollment. Adverse events were not collected for participants in the standard of care study arm.
Description: Adverse events were limited to TPE-associated complications of: hypotension, hypocalcemia, citrate toxicity, angiotensin-converting enzyme (ACE) inhibitor reactions, transfusion-associated circulatory overload, transfusion-related acute lung injury, transfusion-associated dyspnea, allergic reaction, hypotensive transfusion reaction, febrile non-hemolytic transfusion reaction, acute hemolytic transfusion reaction, delayed hemolytic transfusion reaction, and transfusion-transmitted infection.
Arm/Group | Therapeutic Plasma Exchange (TPE) | Standard of Care
All-Cause Mortality (participants affected / at risk) | 2/10 | 5/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/0
Other Adverse Events (participants affected / at risk) | 1/10 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Therapeutic Plasma Exchange (TPE) (N=10) | Standard of Care (N=0)
Mild tachycardia (Cardiac disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/96/NCT04441996/Prot_SAP_000.pdf